CLINICAL TRIAL: NCT04888520
Title: Strength and Muscle Activation of Runners Quadriceps After Eight Weeks of Intervention With Elastic Bandage - A Randomized Controlled Clinical Trial
Brief Title: Strength and Muscle Activation of Runners Quadriceps After 8 Weeks of Intervention With Elastic Bandage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rodrigo Antonio Carvalho Andraus (Other)
Responsible Party: Sponsor-Investigator, Rodrigo Antonio Carvalho Andraus, Coordinator of Stricto Sensu Program in Rehabilitation Sciences, Universidade Norte do Paraná
Organization: Universidade Norte do Paraná (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3.059.113: Projeto Marieli
Record Dates: First submitted 2021-01-06; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-04

CONDITIONS: Muscle Strength
Keywords: Muscle strength; Peak Torque; Electromyography; Athletes
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: The muscle strength of the right knee flexors and extensors will be verified using the isokinetic dynamometer and the muscular activation of the right knee extensors (rectus femoris muscle) will be assessed using surface electromyography. The elastic bandage will be applied over the muscular belly of the right rectus femoris muscle. Initially, all participants will be evaluated without tape, immediately receiving it without tension and, after 20 minutes of rest, they will be reassessed. All will be randomized into two groups and both will receive adhesive tape with or without tension in the application. In the eighth and last week, before the last application of the tape, everyone will be reevaluated without the tape. Then, the last application of the adhesive tape will be carried out with or without tension (according to their respective groups) and after 20 minutes of rest, everyone will be evaluated again with the last application of the tape.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All participants will receive the intervention (application of elastic bandage) and will be blind to which of the two groups belongs. All interventions will be carried out in a private room, one participant at a time. The evaluators (initial and final) and the researcher responsible for analyzing the results will also be blind to the conditions of the groups analyzed. However, the professional who applies the intervention will have knowledge of which group each participant belongs to based on the process of randomizing the participants into two groups. Randomization will be performed by a collaborator not involved in the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tensioning protocol of the elastic bandage (WT) (Experimental): The group will have progressive tension throughout the week - based on the reduction of the tape in relation to the size of the applied area (which will always be the same), which generates a longitudinal tension of the tape in relation to the participant's skin. The Therapy Tex® brand has the elastic deformation capability of up to 40%. The tensioning protocol of the elastic bandage will work with 20% of the elastic deformation capacity of the bandage. The tension will be given from point A to point B in order to generate excitatory stimuli. The percentage of 20% reduction in tension will be distributed over the 7 weeks of intervention, and the first week of the protocol included application without tension. The tape reduction will be controlled by the formula: (size of the application area on the skin*20% /7 weeks= size of the tape to be cut in each of the 7 applications starting from the second week. Tape size and tape application area will be calculated in centimeters (cm).
  Interventions: Device: Adhesive elastic bandage
- Free tension (Placebo Comparator): The group will have no tension in any of its tape applications; that way the size of the tape over the applied area will always be the same.
  Interventions: Device: Adhesive elastic bandage

INTERVENTIONS:
Device: Adhesive elastic bandage — The base of the tape should be applied 5 cm below the origin of the rectus femoris (lower anterior iliac spine), going towards its insertion (base of the patella, through supra-patellar ligament), without tension in this part of the tape (2 to 3 cm initial) in order to avoid discomfort. The application mode will be in "I" ("I-strip"). The participants will be in the supine position, with the hip flexed at 30° and the knee flexed at 60°. The applications of the tape will be carried out every Monday, before the first day of running training of the week and should remain until Friday, when it will be removed by the researcher after the last day of running training of the week. If the elastic bandage unstuck alone from the skin before this period, the event should be immediately reported to the therapist.
  Other Names: Kinesio Tape; Kinesio Taping; Kinesiotape; Kinesiotaping; Functional elastic bandage

SUMMARY:
It is a controlled and randomized clinical trial with the objective of verifying the acute and chronic effects (8 weeks) of elastic banding in runners. Thus, we have as hypotheses of this research: The elastic bandage indirectly influences the muscular strength to the extent that it supposedly can alter the muscular activation verified through the surface electromyography in individuals submitted to the training as the running training. The elastic bandage has clinical significance, however, it does not present statistical significance on muscle strength and activation in individuals submitted to training as running training. To confirm these hypotheses, the muscle strength of the flexors and extensors of the right knee will be checked by means of the isokinetic dynamometer and the muscular activation of the extensors of the right knee (rectus femoris muscle) will be assessed by means of surface electromyography. The elastic bandage will be applied according to a specific protocol in "I" over the muscular belly of the right femoral rectus muscle (which will be submitted to evaluations). All participants will be evaluated without applying adhesive tape and will receive the first application of the tape without tension. Then, after 20 minutes of rest, they will be reassessed with the tape. Participants will be randomized into two groups and both will receive the adhesive tape (with or without tension according to randomization). Then the evaluations will be repeated (all will be reevaluated without the tape and with the tape (with or without tension according to the protocol).

DETAILED DESCRIPTION:
It is a controlled and randomized clinical trial in order to verify the acute and chronic effects (8 weeks of application) of the elastic bandage in runners. hus, we have as hypotheses of this research: The elastic bandage indirectly influences the muscular strength to the extent that it supposedly can alter the muscular activation verified through the surface electromyography in individuals submitted to the training as the running training. The elastic bandage has clinical significance, however, it does not present statistical significance on muscle strength and activation in individuals submitted to training as running training. To confirm these hypotheses, the muscle strength of the flexors and extensors of the right knee will be checked by means of the isokinetic dynamometer and the muscular activation of the extensors of the right knee (rectus femoris muscle) will be assessed by means of surface electromyography. The elastic bandage will be applied according to a specific protocol in "I" over the muscular belly of the right femoral rectus muscle (which will be submitted to evaluations). Initially all participants will be evaluated without applying adhesive tape and, in sequence, they will receive the first application of the tape (for all participants, the tape will be applied without tension) and after 20 minutes of rest, they will be reassessed with the application of the adhesive tape . After the initial assessment, participants will be randomized into two groups and both will receive adhesive tape. The FT (free tension) group will have no tension in any of its tape applications; and the WT (with tension) group will have progressive tension over 8 weeks of intervention (with reduction of the tape length over the weeks, in relation to the same size of the applied area, which generates a longitudinal tension of the tape in relation to skin of the participant). In the eighth and last week of intervention, before the last application of the tape, everyone will be evaluated again (strength and muscle activation) without the tape. Then, the last application of the tape will be performed with or without tension (according to their respective groups) and after 20 minutes of rest, the evaluation of all participants will be performed again with the last application of the tape to the rectus femoris muscle.

ELIGIBILITY:
Inclusion Criteria:

1. being between 18 and 60 years old;
2. being physically able to participate in the experimental study;
3. being completely independent in carrying out basic activities of daily living;
4. not having a physical, hearing or visual impairment that prevents the exams from being performed or making use of prostheses or orthopedic orthoses;
5. having no history of injury to the knee, ankle or hip;
6. has no allergy to elastic bandages;
7. having time to participate in the interventions;
8. has no cognitive impairment according to the Mini Mental State Examination (MMSE);
9. has a training frequency of at least twice a week for more than three months.

Exclusion Criteria:

1. Participants who fail to complete evaluations and/or interventions for any reason
2. Participants who, for some reason, decide to withdraw consent for the research will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in muscle strength of the rectus femoris muscle after 8 weeks of application of the elastic bandage | Initial evaluation will be followed by 8 weeks of intervention with the use of elastic bandage and in the last week the reevaluation will be carried out.
  The dynamometer must be properly calibrated and the evaluation will be carried out with the participant seated and stabilized in the chair with a hip flexion of 85°, with a belt positioned horizontally in the pelvic region and two crossed belts in front of the trunk, in the thoracic region, while another belt will stabilize the thigh of the lower limb contralateral to the evaluated limb. The equipment's rotation axis must be aligned parallel to the axis of the evaluated knee joint (lateral epicondyle), and the lower limb will be fixed to the dynamometer lever arm, with the support pad two centimeters from the heel. The participant will have a brief familiarization with the equipment. They will have visual feedback on the monitor screen. 4 evaluation moments: 2 initial (without elastic bandage; and with elastic bandage, but without tension applied to the elastic bandage); 2 final (without elastic bandage; and with elastic bandage-with or without tension, according to the randomization)

SECONDARY OUTCOMES:
Changes in activation of the rectus femoris muscle (surface electromyography) after 8 weeks of intervention with elastic bandage | Initial evaluation will be followed by 8 weeks of intervention with the use of elastic bandage and in the last week the reevaluation will be carried out.
  The skin must be free of hair and clean with a cotton soaked in 70% alcohol to decrease the impedance of the area, preparing it for the placement of the electrodes. The electrodes will be positioned bilaterally in relation to the orientation of the muscle fibers of the rectus femoris muscle. The EMG signal will be captured with 2 bipolar electrodes and filtered through a bandpass between 25 and 450Hz with a sampling frequency of 2000Hz. With a low frequency filter of 20Hz, a high frequency filter of 1,000Hz and a common mode rejection rate of more than 110dB. The reference electrode will be positioned in the spinous process of the vertebral level C7. Normalization of EMG = Maximum Voluntary Isometric Contraction. 4 evaluation moments: 2 initial (without elastic bandage; and with elastic bandage, but without tension applied to the elastic bandage); 2 final (without elastic bandage; and with elastic bandage-with or without tension, according to the randomization).

CONTACTS AND LOCATIONS:
Overall Officials: Marieli R Stocco, PhD Student, Principal Investigator

IPD SHARING:
Plan to Share IPD: No
There is no need for a plan to make IPD available.

DOCUMENTS (1):
  • Informed Consent Form (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT04888520/ICF_000.pdf